CLINICAL TRIAL: NCT01493440
Title: Atosiban Improves Implantation and Pregnancy Rates in Patients With Repeated Implantation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: An Sinh Hospital (Other)
Collaborators: Vietnam National University (Other)
Responsible Party: Principal Investigator, Vuong Thi Ngoc Lan, Lecturer and Researcher, Department of Obstetrics and Gynecology, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVFAS1103
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Repeated Implantation Failure
Keywords: atosiban; clinical pregnancy; implantation rate; uterine contractility; IVF-ET
MeSH Terms: interventions — atosiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atosiban (Other)
  Interventions: Drug: atosiban

INTERVENTIONS:
Drug: atosiban — Atosiban was administered as a 6.75mg IV bolus dose 30 minutes prior to embryo transfer followed by a 1-hour IV infusion at dose of 18 mg/h then a 2-hour IV infusion at 6 mg/h.
  Other Names: Tractocile

SUMMARY:
Atosiban, administered at embryo transfer, can improve the implantation rate and the clinical pregnancy rate in patients with repeated implantation failure undergoing IVF-ET (in-vitro fertilization and embryo transfer).

DETAILED DESCRIPTION:
Atosiban is a mixed oxytocin and vasopressin V1A receptor antagonist.Combined antagonism at oxytocin and vasopressin V1A receptors reduces uterine contractions with a corresponding decrease in intrauterine production of prostaglandin F2alpha and improved uterine blood supply. These effects are of potential benefit for implantation support during IVF-ET cycles.

ELIGIBILITY:
Inclusion Criteria:

* had repeated implantation failure
* have at least 1 good quality embryo for transfer

Exclusion Criteria:

* uterine abnormalities that could compromise the implantation process (e.g. fibroids, endometrial polyp, bicornuate uterus, adhesion of uterine cavity)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 5 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lan TN Vuong, MD, Principal Investigator — University of Medicine and Pharmacy of Ho Chi Minh City
Locations (1):
- IVFAS, An Sinh Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

REFERENCES:
- [Background] Moraloglu O, Tonguc E, Var T, Zeyrek T, Batioglu S. Treatment with oxytocin antagonists before embryo transfer may increase implantation rates after IVF. Reprod Biomed Online. 2010 Sep;21(3):338-43. doi: 10.1016/j.rbmo.2010.04.009. Epub 2010 Apr 18. PMID 20638340